CLINICAL TRIAL: NCT02661542
Title: A Phase 1/2a, Dose-escalation Study of FF-10502-01 for the Treatment of Advanced Solid Tumors and Lymphomas
Brief Title: Study of FF-10502-01 in Patients With Advanced Solid Tumors and Lymphomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fujifilm Pharmaceuticals U.S.A., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FF1050201US101
Record Dates: First submitted 2016-01-13; First posted 2016-01-22 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Solid Tumors; Lymphomas
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Phase 1: Lowest dose of FF-10502-01 (Experimental): FF-10502-01 will be administered intravenously (IV) on Days 1, 8, and 15 of a 28 day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
  Interventions: Drug: FF-10502-01
- Phase 1: 1.5x lowest dose of FF-10502-01 (Experimental): FF-10502-01 will be administered intravenously (IV) on Days 1, 8, and 15 of a 28 day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
  Interventions: Drug: FF-10502-01
- Phase 1: 2.25x lowest dose of FF-10502-01 (Experimental): FF-10502-01 will be administered intravenously (IV) on Days 1, 8, and 15 of a 28 day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
  Interventions: Drug: FF-10502-01
- Phase 1: 3.375x lowest dose of FF-10502-01 (Experimental): FF-10502-01 will be administered intravenously (IV) on Days 1, 8, and 15 of a 28 day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
  Interventions: Drug: FF-10502-01
- Phase 1: 5x lowest dose of FF-10502-01 (Experimental): FF-10502-01 will be administered intravenously (IV) on Days 1, 8, and 15 of a 28 day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
  Interventions: Drug: FF-10502-01
- Phase 1: 7.5x lowest dose of FF-10502-01 (Experimental): FF-10502-01 will be administered intravenously (IV) on Days 1, 8, and 15 of a 28 day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
  Interventions: Drug: FF-10502-01
- Phase 1: 11.25x lowest dose of FF-10502-01 (Experimental): FF-10502-01 will be administered intravenously (IV) on Days 1, 8, and 15 of a 28 day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
  Interventions: Drug: FF-10502-01
- Phase 1: 16.875x lowest dose of FF-10502-01 (Experimental): FF-10502-01 will be administered intravenously (IV) on Days 1, 8, and 15 of a 28 day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
  Interventions: Drug: FF-10502-01
- Phase 1: 25x lowest dose of FF-10502-01 (Experimental): FF-10502-01 will be administered intravenously (IV) on Days 1, 8, and 15 of a 28 day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
  Interventions: Drug: FF-10502-01
- Phase 2a: FF-10502-01 at MTD in Pancreatic Cancer (Experimental): FF-10502-01 will be administered intravenously (IV) on Days 1, 8, and 15 of a 28 day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
  Interventions: Drug: FF-10502-01
- Phase 2a: FF-10502-01 at MTD in Solid Tumors (Experimental): FF-10502-01 will be administered intravenously (IV) on Days 1, 8, and 15 of a 28 day cycle. The dose-escalation will proceed until Maximum Tolerated Dose (MTD) is reached. The treatment will continue until disease progression, intolerable toxicity or investigation/subject decision.
  Interventions: Drug: FF-10502-01

INTERVENTIONS:
Drug: FF-10502-01

SUMMARY:
A Phase 1/2a, dose-escalation study of FF-10502-01 in Patients with Advanced Solid Tumors and Lymphomas. A total of up to 9 cohorts will be enrolled in Phase 1 to establish the MTD. Phase 2 will consist of 2 cohorts: Cohort 1 will include subjects with Pancreatic Cancer. Cohort 2 will include subjects with another tumor type enrolled in the Phase 1 dose-escalation phase who have demonstrated Clinical Benefit by Week 16.

DETAILED DESCRIPTION:
Subjects will receive doses of FF-10502-01 intravenously (IV) weekly for three weeks, repeated every 28 days (= 1 cycle). Disease assessments, based on computed tomography (CT), magnetic resonance image (MRI), and, for lymphoma, [18F]-fluorodeoxyglucose positron emission tomography (FDG-PET) scans, will be obtained at Week 8 and every 8 weeks thereafter until documented progression of disease (PD). Subjects who demonstrate clinical benefit will be allowed to continue therapy with FF-10502-01 until progression of disease, observation of unacceptable adverse events, intercurrent illness or changes in the subject's condition that prevents further study participation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Histologically or cytologically confirmed advanced or metastatic solid tumor or l lymphoma, that is refractory to standard therapy, relapsed after standard therapy, or for which no standard therapy available that is expected to improve survival by at least three months
* At least 4 weeks beyond the last chemotherapy (or ≥ 5 half-lives for targeted agents, whichever is shorter), radiotherapy, major surgery or experimental treatment and recovered from all acute toxicities (≤ Grade 1)
* Adequate performance status: Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Life expectancy of ≥ 3 months
* Adequate hematologic parameters without ongoing transfusional support:
* Hemoglobin (Hb) ≥ 9 g/dL
* Absolute neutrophil count (ANC) ≥ 1.0 x 109 cells/L
* Platelets ≥ 100 x 109 cells/L
* Adequate renal and hepatic function:
* Creatinine ≤ 1.5 x the upper limit of normal (ULN), or calculated creatinine clearance ≥ 60 mL/minute x 1.73 m2 per the Cockcroft-Gault formula
* Total bilirubin ≤ 2 times the upper limit of normal (ULN) unless due to Gilbert's disease
* ALT/AST ≤ 2.5 times ULN, or < 5 times ULN for subjects with liver metastases
* QT interval corrected for rate (QTc) ≤ 480 msec on the electrocardiogram (ECG) obtained at Screening
* Negative serum pregnancy test within 14 days prior to the first dose of study therapy for women of child-bearing potential (WCBP), defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally post-menopausal for at least 24 consecutive months (i.e., who has had menses any time in the preceding 24 consecutive months). Sexually active WCBP and male subjects must agree to use adequate methods to avoid pregnancy (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study and for 28 days after the completion of study treatment.
* Ability to provide written informed consent

Exclusion Criteria:

* Serious cardiac condition within the last 6 months, such as uncontrolled arrhythmia, myocardial infarction, unstable angina or heart disease defined by the New York Heart Association (NYHA) Class III or Class IV
* Concomitant medication(s) that may cause QTc prolongation or induce Torsades de Pointes, with the exception of anti-microbials that are used as standard of care to prevent or treat infections and other such drugs that are considered by the Investigator to be essential for patient care
* Active central nervous system (CNS) malignant disease in subjects with a history of CNS malignancy. Subjects with stable, prior or currently treated brain metastases are allowed.
* Known positive for human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV)
* Active infection requiring intravenous (IV) antibiotic usage within the last week prior to study treatment
* Any other medical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence to study requirements or confound the interpretation of study results
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (Safety and Tolerability) | 33 Months
  Safety and tolerability assessed by adverse events (AEs), and serious adverse events. (SAEs)

SECONDARY OUTCOMES:
Determination of overall response rates | Responses assessed at end of C2 and every 2 cycles thereafter through 6 months following last dose of study drug (every 28 days=1 cycle).
  Determination of overall response rates
Determination of duration of response. | Assessed at end of C2 and every 2 cycles thereafter through 6 months following last dose of study drug
  duration of response is determined
Determination of duration of stable disease (SD) as measured from time of 1st evidence of response to time of 1st evidence of progressive disease as measured by CT or MRI. | Assessed at end of C2 and every 2 cycles thereafter through 6 months following last dose of study drug
  measurement of stable disease
Evaluate progression-free survival (PFS) | Responses and survival assessed, at the end of C2 and every 2 cycles thereafter through 6 months following last dose of study drug
  measurement of PFS
Evaluate overall survival (OS) | Assessed by telephone call at end of C2 and every 2 cycles thereafter through 6 months following last dose of study drug
  measurement of OSS
Evaluate the mean plasma concentrations of FF-10502-01 | Assessed at Cycle 1 Day 1, and Cycle 1 Day 15
  measurement of plasma concentrations
Evaluate FF-10502-01 incorporation into whole blood cellular DNA by LC-MS/MS as a pharmacodynamic marker | Assessed at Cycle 1 Day 1, Cycle 1 Day , Cycle 1 Day 15, Cycle 1, Day 22, Cycle 2 Day 1, at the end of Cycle 2 and ever 2 cycles thereafter up to 24 weeks.
  measurement of cellular DNA

CONTACTS AND LOCATIONS:
Overall Officials: Filip Janku, MD, Principal Investigator — University of Texas MD Anderson Center; Gerald Falchook, MD, Principal Investigator — Sarah Cannon Research Institute-Denver
Locations (2):
- United States (2):
  - Sarah Cannon Research Institute at HealthOne, Denver, Colorado
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No